CLINICAL TRIAL: NCT00971659
Title: Acute Effect of a GLP-1-Analogue (Exenatide) and of a DPP-4-Inhibitor (Sitagliptin) in Subjects With Type 2 Diabetes Treated With Insulin Glargine Once Daily
Brief Title: Adjunctive Therapy of Exenatide or Sitagliptin to Insulin Glargine in Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Profil Institut für Stoffwechselforschung GmbH (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Christoph Kapitza, MD, Profil Institut für Stoffwechselforschung GmbH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 49/0316-Adjunct
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2009-09-04 (Estimated); Status verified 2009-09

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Exenatide; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- insulin glargine + exenatide + metformin (Experimental)
  Interventions: Drug: insulin glargine + exenatide + preexisting metformin
- Insulin glargine + sitagliptin + metformin (Experimental)
  Interventions: Drug: insulin glargine + sitagliptin + preexisting metformin
- insulin glargine + metformin (Active Comparator)
  Interventions: Drug: insulin glargine + preexisting metformin

INTERVENTIONS:
Drug: insulin glargine + exenatide + preexisting metformin — insulin glargine once daily subcutaneously over 4 weeks, dose adjustment according to a treat-to-target algorithm, exenatide 5ug twice daily subcutaneously for 2 weeks, then 10ug twice daily for 2 weeks, continuation of preexisting metformin
  Other Names: Lantus; Byetta
  Arms: insulin glargine + exenatide + metformin
Drug: insulin glargine + sitagliptin + preexisting metformin — insulin glargine once daily subcutaneously over 4 weeks, dose adjustment according to a treat-to-target algorithm, sitagliptin 100 mg once daily in the morning over 4 weeks, continuation of preexisting metformin
  Other Names: Lantus; Januvia
  Arms: Insulin glargine + sitagliptin + metformin
Drug: insulin glargine + preexisting metformin — insulin glargine once daily subcutaneously over 4 weeks, continuation of preexisting metformin
  Other Names: Lantus
  Arms: insulin glargine + metformin

SUMMARY:
This study investigated a 4-week adjunctive therapy of either a GLP-1 analog (exenatide), or a DPP-4 inhibitor (sitagliptin), given to a basal insulin analog (insulin glargine), and their effect on blood glucose control, versus insulin glargine alone as active comparator in type 2 diabetes.

DETAILED DESCRIPTION:
Due to the different mechanisms of action of the long-acting insulin analog insulin glargine and both a GLP-1 analog (exenatide) and a DPP-4-inhibitor (sitagliptin), it could be a promising approach to combine insulin glargine with either exenatide or sitagliptin for optimum control of fasting and postprandial blood glucose values. Thus, in the present study the influence of either exenatide or sitagliptin as a 4-week adjunctive therapy to a basal insulin (insulin glargine) was investigated versus insulin glargine alone as active comparator in subjects with type 2 diabetes. Preexisting metformin was continued, sulfonylureas, if any, were stopped. In particular, the effects on postprandial blood glucose excursion following ingestion of a standard breakfast, assessed after 4 weeks of treatment, the effects on mean daily blood glucose, on self-measured 7-point profiles, the percentage of subjects reaching ADA treatment goals (HbA1c < 7.0%) at the end of treatment, on fasting lipid profile, on HOMA index, weight, hypoglycemic episodes and general safety were assessed. The study consisted of a screening visit, a 4-8 week (depending on pre-treatment) run-in period, a 4-week treatment period, and a follow-up visit. There were weekly visits at the site and twice weekly telephone contacts.

ELIGIBILITY:
Inclusion Criteria:

* male or female subjects aged between 35 and 70 years, inclusive
* type 2 diabetes with duration >6 months and <10 years
* for at least 3 months: treatment solely with a long- or intermediate-acting insulin formulation (insulin glargine, insulin detemir, or NPH insulin) with or without a stable dose of metformin or treatment solely with a stable dose of metformin or combination of stable doses of metformin plus sulfonylureas
* HbA1c >=7.0% and <=10.0%
* if treated with antihypertensive or lipid lowering agents, the treatment regimen had to be stable during 3 months prior to study start
* written informed consent

Exclusion Criteria:

* history or presence of cancer or any clinically relevant diseases
* chronic heart failure NYHA class III or IV, unstable angina pectoris or myocardial infarction within the previous 6 months
* recurrent hypoglycemia
* abnormal lab tests at screening (ALAT and/or ASAT >=3 times ULN), creatinine >1.6 mg/dL in males and >1.4 mg/dL in females
* clinically relevant ECG findings at screening
* treatment with a rapid-acting insulin or with a mixed insulin formulation during the previous 3 months
* treatment with any other OHA than metformin or metformin plus sulfonylureas during the previous 3 months
* any systemic or topical treatment with drugs known to influence glucose metabolism

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-01; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
the unadjusted 6-hour postprandial blood glucose excursion (AUCBG0-6h) following ingestion of a standardized breakfast | after 4 weeks of treatment

SECONDARY OUTCOMES:
mean daily blood glucose (BG) from 7-point 24h BG profiles, fasting BG, self-measured 7-point BG profiles, percentage of subjects achieving ADA HbA1c treatment goals, fasting lipid profiles, HOMA-IR index, hypoglycemic episodes | after 4 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Arnolds, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

REFERENCES:
- [Derived] Arnolds S, Dellweg S, Clair J, Dain MP, Nauck MA, Rave K, Kapitza C. Further improvement in postprandial glucose control with addition of exenatide or sitagliptin to combination therapy with insulin glargine and metformin: a proof-of-concept study. Diabetes Care. 2010 Jul;33(7):1509-15. doi: 10.2337/dc09-2191. Epub 2010 Mar 31. PMID 20357372